CLINICAL TRIAL: NCT00763568
Title: Study of a 4-Week Lead-In With Nitazoxanide Followed By 36 Weeks of Nitazoxanide Plus Peginterferon Alfa-2a in the Treatment of Chronic Hepatitis C
Brief Title: 4-Week Lead-In With Nitazoxanide Followed by 36 Weeks Nitazoxanide and Peginterferon Alfa-2a in Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Romark Laboratories, L.C., Romark Laboratories, L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM01-3037
Record Dates: First submitted 2008-09-26; First posted 2008-10-01 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Viral hepatitis
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — nitazoxanide; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitazoxanide (Experimental): One nitazoxanide 500 mg tablet orally twice a day for 4 weeks followed by one nitazoxanide 500 mg tablet orally twice a day plus weekly injections of 180µg peginterferon alfa-2a for 36 weeks.
  Interventions: Drug: Nitazoxanide; Biological: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Nitazoxanide — One nitazoxanide 500 mg tablet orally twice a day for 4 weeks followed by one nitazoxanide 500 mg tablet orally twice a day plus weekly injections of 180µg peginterferon alfa-2a for 36 weeks.
  Other Names: Alinia
Biological: Peginterferon alfa-2a — One nitazoxanide 500 mg tablet orally twice a day for 4 weeks followed by one nitazoxanide 500 mg tablet orally twice a day plus weekly injections of 180µg peginterferon alfa-2a for 36 weeks.
  Other Names: PEGASYS

SUMMARY:
The purpose of this study is to determine if taking nitazoxanide alone for 4 weeks followed by 36 weeks of nitazoxanide plus peginterferon is superior to peginterferon plus ribavirin (standard of care) for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C

Exclusion Criteria:

* Previously failed to respond to at least 12 weeks of peginterferon plus ribavirin combination therapy.
* Unable to take oral medication.
* Females who are either pregnant, breast-feeding or not using birth control.
* Males whose female partners are pregnant or plan to become pregnant.
* Other causes of liver disease (for example, autoimmune hepatitis, decompensated liver disease).
* Patients with HIV, HAV, HBV or HDV.
* Patients with a history of alcoholism or with an alcohol consumption of more than 40 grams per day.
* Patients with hemoglobinopathies (for example, thalassemia major, sickle-cell anemia).
* History of hypersensitivity or intolerance to nitazoxanide or peginterferon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response | 24 weeks after the end of treatment

SECONDARY OUTCOMES:
End of treatment virologic response | At the end of treatment
Early virologic response | After 12 weeks of combination therapy
Rapid virologic response | After 4 weeks of combination therapy
ALT normalization | 24 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Asem Elfert, MD, Principal Investigator — Tanta University School of Medicine
Locations (1):
- Digestive Disease Center, Tanta, Egypt